CLINICAL TRIAL: NCT05840718
Title: Impact of Thiamine Supplementation on Clinical Outcomes of Patients With Septic Shock: a Retrospective Before-after Study
Brief Title: Supplemental Thiamine in Septic Shock: A Before-after Study
Status: Completed | Type: Observational
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, Clinical Professor, Hospital Sao Domingos
Other Study IDs: 13/2023
Record Dates: First submitted 2023-04-16; First posted 2023-05-03 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Septic Shock
Keywords: Septic shock; Thiamin; Critically ill patients; Mortality; Surviving sepsis campaign
MeSH Terms: conditions — Shock, Septic | interventions — Thiamine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Septic shock patients treated according surviving sepsis campaign 2021 guidelines
- Intervention group: Septic shock patients treated according surviving sepsis campaign 2021 guidelines supplemented with thiamin 200 mg in 50 ml 5% dextrose twice daily for 7 days.
  Interventions: Drug: Thiamin

INTERVENTIONS:
Drug: Thiamin — Patients in thiamine group received two daily dosis of 200 mg of thiamin diluted in 50 ml of 5% dextrose during 7 days
  Groups: Intervention group

SUMMARY:
This controlled before-and-after study analyse the impact of thiamine supplementation on outcomes of patients with septic shock treated according to the surviving sepsis campaign 2021 guidelines

DETAILED DESCRIPTION:
Vitamin B1 (Thiamine) is a water-soluble vitamin that plays an important role in various biological processes. The active form is thiamine pyrophosphate, an essential cofactor in enzyme systems involved in carbohydrate metabolism and energy production. Recently, the role of thiamine in critically ill patients has gained prominence and septic shock has deserved special attention (1,2). It is important to emphasize that in these situations the clinical syndromes have low sensitivity and specificity for clinical diagnosis, which means that a high level of suspicion must be exercised in these situations. Donnino et al (3) analyzed 88 patients with septic shock in a prospective, randomized, double-blind study. The study showed that the administration of thiamine at a dose of 200 mg every 12 hours for 7 days had a significant impact on mortality only in patients who had reduced serum levels of thiamine. Woolum et al (4 ) retrospectively analyzed the impact of a single dose of Thiamine administered in the 24 hours that preceded the diagnosis of septic shock and compared with patients who did not receive the vitamin and identified improvement in lactate clearance and reduction in 28-day mortality in the thiamine group. Petsakul et al (5) evaluated the effect of thiamine administration in patients with septic shock and need for vasopressors and showed a significant reduction in the vasopressor dose in addition to improvement in lactate clearance. A recent meta-analysis including 5 studies and 645 patients with septic shock analyzed the impact of thiamine use on mortality. The study included 3 prospective randomized studies and 2 retrospective observational studies. The result showed a borderline beneficial effect on mortality. Regarding to HAT (Hydrocortisone, ascorbic acid and thiamine) therapy after the initial study by Marik et al. (7 ) at least 3 prospective randomized studies failed to repeat the good results of the initial study (8,9,10).

The sepsis management protocol at the São Domingos hospital underwent important changes from December 2021 to October 2022. In December, changes were incorporated in the protocol based on the new version of the Surviving Sepsis Campaign 2021 that had been launched the previous month ( 11). In April 2022 the SOSD (salvage, optimization, stabilization and de-resuscitation) systematics (12) was incoporated in the management of septic shock and in October 2022 thiamine use was implemented. Thiamine was incorporated into the protocol, although there are still no robust studies to indicate its use because, despite the implementation of previous measures with exceptional results in sepsis, between January and September 2022, mortality from sepsis was 1.69%, in the septic shock we had evolved little or nothing with mortality in the same period of 70%. In October, thiamine was started in isolated cases and as of November 2022, the investigators started using thiamine systematically and in all cases of septic shock at a dose of 200 mg EV every 12 hours for 7 days. In this controlled before-and-after study, the investigators compared outcomes of patients treated for septic shock between November 2022 and March 2023 with patients diagnosed with septic shock treated between May and September 2022.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* presence of documented or suspected infection, SOFA score ≥ 2, serum lactate levels > 18 mg/dL and hypotension, MAP < 65 mm Hg maintained after volume expansion of at least 30 ml/kg in the first 2 hours of treatment followed by noradrenaline vasopressor dependence (with or without vasopressin) during the first 6 hours of treatment.

Exclusion Criteria:

* pregnant women
* patients treated only with comfort measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a retrospective before-after study. Included were all patients with inclusion criteria admitted to a 13-bed surgical ICU, a 12-bed medical and a 12-bed high-complexity surgical and trauma ICU .during the 2 study periods: May 1 to September 30, 2022, control group and November 1, 2022 to March 31, 2023, study group.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Compare lactate clearance between intervention (thiamine supplemented) and control group. | 30 days
  Lactate clearance defined as a consistent serum lactate level below 19 mg/dL after the start of treatment for septic shock

SECONDARY OUTCOMES:
Comparison of mortality rate between intervention (thiamine supplemented) and control | 30 days
  To determine the mortality rate of patients with septic shock who received thiamine supplementation 200 mg twice daily for 7 days (intervention group) compared to a group that did not receive thiamine. Both groups treated according to Surviving Sepsis Campaign guidelines version 2021.
Comparison of vasopressor-free days during ICU stay between the groups intervention and control | 30 days
  Compare the vasopressor-free days between the two groups during the ICU stay
Comparison of vantilation-free days during ICU stay between the groups intervention and control | 30 days
  Compare ventilation-free days between the two groups during the ICU stay
Compare the use of renal replacement therapy, n (%), initiated after 48 hours of septic shock between the groups intervention (thiamine supplementation) and control group | 30 days
  - Compare the use of renal replacement therapy initiated after 48 hours of septic shock between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: ISNARA S CARVALHO, RN, Principal Investigator — Hospital Sao Domingos
Locations (2):
- Brazil (2):
  - Hospital Sao Domingos, São Luís, Maranhão
  - Hospital São Domingos, São Luís, Maranhão

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cruickshank AM, Telfer AB, Shenkin A. Thiamine deficiency in the critically ill. Intensive Care Med. 1988;14(4):384-7. doi: 10.1007/BF00262893. PMID 3136196
- [Result] Costa NA, Gut AL, de Souza Dorna M, Pimentel JA, Cozzolino SM, Azevedo PS, Fernandes AA, Zornoff LA, de Paiva SA, Minicucci MF. Serum thiamine concentration and oxidative stress as predictors of mortality in patients with septic shock. J Crit Care. 2014 Apr;29(2):249-52. doi: 10.1016/j.jcrc.2013.12.004. Epub 2013 Dec 14. PMID 24412011
- [Result] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Result] Woolum JA, Abner EL, Kelly A, Thompson Bastin ML, Morris PE, Flannery AH. Effect of Thiamine Administration on Lactate Clearance and Mortality in Patients With Septic Shock. Crit Care Med. 2018 Nov;46(11):1747-1752. doi: 10.1097/CCM.0000000000003311. PMID 30028362
- [Result] Petsakul S, Morakul S, Tangsujaritvijit V, Kunawut P, Singhatas P, Sanguanwit P. Effects of thiamine on vasopressor requirements in patients with septic shock: a prospective randomized controlled trial. BMC Anesthesiol. 2020 Nov 9;20(1):280. doi: 10.1186/s12871-020-01195-4. PMID 33167911
- [Result] Kanchanasurakit S, Suthumpoung P, Santimaleeworagun W, Nakaranurack C, Huynh NS, Srisawat C, Nunta M, Chirakan V, Saokaew S. Effectiveness of thiamine therapy in mortality rate in patients with septic shock: A systematic review and meta-analysis. Int J Crit Illn Inj Sci. 2021 Apr-Jun;11(2):86-94. doi: 10.4103/IJCIIS.IJCIIS_159_20. Epub 2021 Jun 29. PMID 34395210
- [Result] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Result] Fujii T, Luethi N, Young PJ, Frei DR, Eastwood GM, French CJ, Deane AM, Shehabi Y, Hajjar LA, Oliveira G, Udy AA, Orford N, Edney SJ, Hunt AL, Judd HL, Bitker L, Cioccari L, Naorungroj T, Yanase F, Bates S, McGain F, Hudson EP, Al-Bassam W, Dwivedi DB, Peppin C, McCracken P, Orosz J, Bailey M, Bellomo R; VITAMINS Trial Investigators. Effect of Vitamin C, Hydrocortisone, and Thiamine vs Hydrocortisone Alone on Time Alive and Free of Vasopressor Support Among Patients With Septic Shock: The VITAMINS Randomized Clinical Trial. JAMA. 2020 Feb 4;323(5):423-431. doi: 10.1001/jama.2019.22176. PMID 31950979
- [Result] Moskowitz A, Huang DT, Hou PC, Gong J, Doshi PB, Grossestreuer AV, Andersen LW, Ngo L, Sherwin RL, Berg KM, Chase M, Cocchi MN, McCannon JB, Hershey M, Hilewitz A, Korotun M, Becker LB, Otero RM, Uduman J, Sen A, Donnino MW; ACTS Clinical Trial Investigators. Effect of Ascorbic Acid, Corticosteroids, and Thiamine on Organ Injury in Septic Shock: The ACTS Randomized Clinical Trial. JAMA. 2020 Aug 18;324(7):642-650. doi: 10.1001/jama.2020.11946. PMID 32809003
- [Result] Sevransky JE, Rothman RE, Hager DN, Bernard GR, Brown SM, Buchman TG, Busse LW, Coopersmith CM, DeWilde C, Ely EW, Eyzaguirre LM, Fowler AA, Gaieski DF, Gong MN, Hall A, Hinson JS, Hooper MH, Kelen GD, Khan A, Levine MA, Lewis RJ, Lindsell CJ, Marlin JS, McGlothlin A, Moore BL, Nugent KL, Nwosu S, Polito CC, Rice TW, Ricketts EP, Rudolph CC, Sanfilippo F, Viele K, Martin GS, Wright DW; VICTAS Investigators. Effect of Vitamin C, Thiamine, and Hydrocortisone on Ventilator- and Vasopressor-Free Days in Patients With Sepsis: The VICTAS Randomized Clinical Trial. JAMA. 2021 Feb 23;325(8):742-750. doi: 10.1001/jama.2020.24505. PMID 33620405
- [Result] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Result] Malbrain MLNG, Martin G, Ostermann M. Everything you need to know about deresuscitation. Intensive Care Med. 2022 Dec;48(12):1781-1786. doi: 10.1007/s00134-022-06761-7. Epub 2022 Aug 6. No abstract available. PMID 35932335